CLINICAL TRIAL: NCT00096993
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy of Pertuzumab (rhuMAb 2C4) in Combination With Gemcitabine and the Effect of Tumor-Based HER2 Activation in Subjects With Platinum-Resistant Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study to Evaluate rhuMab 2C4 and Gemcitabine in Subjects With Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOC3258g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Omnitarg; Cancer; Platinum-Resistant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Gemcitabine; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + gemcitabine (Placebo Comparator): Participants received placebo intravenously on Day 1 of every 3 week cycle for up to 1 year (up to 17 treatment cycles). In addition, participants received gemcitabine 800 mg/m^2 intravenously on Days 1 and 8 of every 3 week cycle for up to 1 year (up to 17 treatment cycles).
  Interventions: Drug: Placebo; Drug: Gemcitabine
- Pertuzumab + gemcitabine (Active Comparator): Participants received pertuzumab intravenously on Day 1 of every 3 week cycle for up to 1 year (up to 17 treatment cycles). Participants received pertuzumab at a loading dose of 840 mg in Cycle 1 followed by a dose of 420 mg in Cycles 2 and beyond. In addition, participants received gemcitabine 800 mg/m^2 intravenously on Days 1 and 8 of every 3 week cycle for up to 1 year (up to 17 treatment cycles
  Interventions: Drug: Gemcitabine; Drug: Pertuzumab

INTERVENTIONS:
Drug: Placebo — Placebo was provided as a single-use formulation for infusion.
  Arms: Placebo + gemcitabine
Drug: Gemcitabine — Gemcitabine was provided as a solution for infusion.
  Other Names: Gemzar
Drug: Pertuzumab — Pertuzumab was provided as a single-use formulation for infusion.
  Other Names: rhuMAb 2C4
  Arms: Pertuzumab + gemcitabine

SUMMARY:
This is a Phase II, randomized, placebo-controlled, double-blind, multicenter clinical trial of pertuzumab in combination with gemcitabine relative to placebo in combination with gemcitabine in subjects with advanced ovarian, primary peritoneal, or fallopian tube cancer that is resistant to platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >= 18 years
* Advanced, histologically documented ovarian, primary peritoneal, or fallopian tube carcinoma
* Representative tumor specimens in paraffin blocks or at least 12 unstained slides with an associated pathology report, obtained at any time prior to entry of study for evaluation of HER2 activation
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension (longest dimension recorded), Or:
* Clinically or radiologically detectable disease (e.g., ascites, peritoneal deposits, mesenteric thickening or lesions that do not fulfill RECIST for measurable disease)
* Platinum-resistant or refractory carcinoma
* Life expectancy >= 12 weeks
* ECOG performance status 0 or 1
* LVEF >= 50%, as determined by ECHO
* Use of an effective means of contraception (for women of childbearing potential)
* Clinical laboratory test results: Granulocyte count >= 1500/uL; Platelet count >= 75,000/uL; Hemoglobin >= 9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbopoeitin [Aranesp(R)] is permitted); Serum bilirubin <= 1.5 the ULN; Alkaline phosphatase, AST, and ALT <= 2.5 ULN (AST, ALT <= 5 ULN for subjects with liver metastasis); Serum creatinine <= 1.5 ULN; International normalized ratio (INR) <= 1.5 and activated partial thromboplastin time (aPTT) <= 1.5 ULN (except for subjects receiving anti-coagulation therapy)

Exclusion Criteria:

* Prior treatment with gemcitabine
* Two or more prior regimens for the treatment of platinum-resistant disease
* Two or more non-platinum-containing regimens for the treatment of platinum-sensitive disease
* Prior treatment with experimental anti-cancer agents within 4 weeks prior to Day 1 (the day the first study treatment infusions are administered)
* Prior treatment with HER2 pathway inhibitors (e.g., Herceptin(R) [trastuzumab], Iressa(R) [gefitinib], Tarceva<TM> [erlotinib hydrochloride], cetuximab, GW572016)
* History or clinical evidence of central nervous system or brain metastases
* Uncontrolled hypercalcemia ( > 11.5 mg/dL)
* Prior exposure of > 360 mg/m^2 doxorubicin or liposomal doxorubicin, > 120 mg/m^2 mitoxantrone, or > 90 mg/m^2 idarubicin
* History of other malignancies within 5 years of Day 1, except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of breast, basal or squamous cell skin cancer
* History of serious systemic disease, unstable angina, myocardial infarction within 6 months prior to Day 1 of treatment, symptoms of CHF, or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia [i.e., atrial fibrillation, paroxysmal supraventricular tachycardia] are eligible)
* Known HIV infection
* Pregnancy or lactation
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1 of treatment
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Patton, M.D., Study Director — Genentech, Inc.
Locations (41):
- United States (41):
  - Univ. of Alabama at Birmingham, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Comp. Cancer Ctr, Berkeley, California
  - California Cancer Crae, Inc, Greenbrae, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Sutter Cancer Center, Sacramento, California
  - Southern California Permanente Medical Group (Kaiser), San Diego, California
  - Sharp Healthcare, San Diego, California
  - Norwalk Medical Group, Norwalk, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Memorial Health Univ. Med. Ctr., Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - University Of Chicago, Chicago, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State Univ. Barbara Ann Karmanos Cancer Inst., Detroit, Michigan
  - Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Cooper Health System, Voorhees Township, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - Ohio State University College of Medicaine, Columbus, Ohio
  - Pelvic Surgery Assoc., Columbus, Ohio
  - Oklahoma Univ. Medical Center, Oklahoma City, Oklahoma
  - Corvallis Clinic, Corvallis, Oregon
  - Kaiser Permanente Northwest Division, Portland, Oregon
  - Womens and Infants Hospital, Providence, Rhode Island
  - Northern Virginia Pelvic Surgery Assoc., Annandale, Virginia
  - Carilion Gyn/Onc, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject in the placebo + gemcitabine arm did not receive any study treatment as the subject died of a cerebrovascular accident prior to the first scheduled dose. This subject was excluded from both the efficacy and safety analyses, per protocol.
Period: Overall Study
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Started | 66 | 65
Completed | 1 | 0
Not Completed | 65 | 65
Not completed — Death | 1 | 0
Not completed — Disease progression | 56 | 53
Not completed — Adverse Event | 2 | 8
Not completed — Subject's decision | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Other unspecified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received any amount of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (11.94) | 57.8 (10.79) | 58.7 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 130
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first day of treatment (Cycle 1, Day 1) to the time of documented disease progression or death, whichever occurred first. Disease progression was assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) was defined as disappearance of all target lesions; Partial Response (PR) was defined as >=30% decrease in the sum of the longest diameter of target lesions and Overall Response (OR) = CR + PR.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Efficacy-evaluable population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Number analyzed (Participants) | 54 | 49
months | 2.6 [1.4 to 3.9] | 2.9 [2.6 to 4.4]

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete or partial response determined on two consecutive occasions ≥ 4 weeks apart. Responses were determined by Response Evaluation Criteria in Solid Tumors (RECIST). A complete response was defined as the disappearance of all target lesions or the disappearance of all non-target lesions and normalization of tumor marker level. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter of target lesions.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Efficacy-evaluable population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Number analyzed (Participants) | 65 | 65
percentage of participants | 4.6 | 13.8

3. Secondary Outcome: Duration of the Objective Response
Description: Duration of the objective response was defined as the time from the initial response to disease progression or death from any cause.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Efficacy-evaluable population: All randomized participants who received at least 1 dose of study medication. Only participants with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Number analyzed (Participants) | 3 | 9
months | NA [4.1 to NA] — Value is not estimable; not reached | 6.9 [4.1 to 7.4]

4. Secondary Outcome: Percentage of Participants Free From Disease Progression at 4 Months
Description: Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to Month 4
Population: Efficacy-evaluable population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Number analyzed (Participants) | 65 | 65
percentage of participants | 37.3 | 47.6

5. Secondary Outcome: Duration of Survival
Description: Duration of survival was defined as the time from randomization until death from any cause.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Efficacy-evaluable population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Number analyzed (Participants) | 65 | 65
months | 13.1 [10.5 to 15.5] | 13.0 [9.6 to 18.5]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the beginning of study treatment until 30 days after discontinuation of study treatment.
Description: Safety population: All participants who received any amount of study treatment.
Arm/Group | Placebo + Gemcitabine | Pertuzumab + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 40/65 | 23/65
Other Adverse Events (participants affected / at risk) | 65/65 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=65) | Pertuzumab + Gemcitabine (N=65)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 8 | 2
VOMITING (Gastrointestinal disorders) | 3 | 1
ILEUS (Gastrointestinal disorders) | 2 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
NAUSEA (Gastrointestinal disorders) | 2 | 0
COLONIC STENOSIS (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 1
CELLULITIS (Infections and infestations) | 1 | 1
INFECTION (Infections and infestations) | 2 | 0
CATHETER RELATED INFECTION (Infections and infestations) | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 2
HYPOTENSION (Vascular disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 1
CATHETER RELATED COMPLICATION (General disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 0
INFUSION RELATED REACTION (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
FEEDING TUBE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Gemcitabine (N=65) | Pertuzumab + Gemcitabine (N=65)
NAUSEA (Gastrointestinal disorders) | 47 | 49
DIARRHOEA (Gastrointestinal disorders) | 39 | 44
VOMITING (Gastrointestinal disorders) | 33 | 32
CONSTIPATION (Gastrointestinal disorders) | 40 | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 26 | 22
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 21 | 12
STOMATITIS (Gastrointestinal disorders) | 11 | 19
DYSPEPSIA (Gastrointestinal disorders) | 13 | 14
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 6
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 10 | 9
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 8 | 5
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 5 | 7
ASCITES (Gastrointestinal disorders) | 9 | 3
DRY MOUTH (Gastrointestinal disorders) | 5 | 2
FLATULENCE (Gastrointestinal disorders) | 3 | 4
ORAL PAIN (Gastrointestinal disorders) | 4 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 4
FATIGUE (General disorders) | 50 | 51
OEDEMA PERIPHERAL (General disorders) | 28 | 20
PYREXIA (General disorders) | 22 | 19
CHILLS (General disorders) | 12 | 12
PAIN (General disorders) | 12 | 12
ASTHENIA (General disorders) | 11 | 7
CHEST PAIN (General disorders) | 7 | 6
MUCOSAL INFLAMMATION (General disorders) | 5 | 7
OEDEMA (General disorders) | 1 | 6
INJECTION SITE PAIN (General disorders) | 5 | 1
INJECTION SITE IRRITATION (General disorders) | 5 | 0
ANAEMIA (Blood and lymphatic system disorders) | 39 | 31
NEUTROPENIA (Blood and lymphatic system disorders) | 29 | 32
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 | 19
LEUKOPENIA (Blood and lymphatic system disorders) | 8 | 9
ANOREXIA (Metabolism and nutrition disorders) | 21 | 18
HYPOKALAEMIA (Metabolism and nutrition disorders) | 20 | 12
DECREASED APPETITE (Metabolism and nutrition disorders) | 15 | 7
DEHYDRATION (Metabolism and nutrition disorders) | 14 | 6
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 13 | 7
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 15 | 5
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 15 | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 15 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 22 | 22
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 23 | 21
HAEMOGLOBIN DECREASED (Investigations) | 10 | 11
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 7 | 8
BLOOD CREATININE INCREASED (Investigations) | 7 | 5
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 | 6
EJECTION FRACTION DECREASED (Investigations) | 7 | 4
NEUTROPHIL COUNT DECREASED (Investigations) | 7 | 3
BLOOD ALBUMIN DECREASED (Investigations) | 5 | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 6 | 3
PLATELET COUNT DECREASED (Investigations) | 7 | 1
WEIGHT DECREASED (Investigations) | 4 | 4
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 4
BLOOD URINE PRESENT (Investigations) | 4 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 | 27
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 9
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 | 5
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 6
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 4
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 20 | 19
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 | 19
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 15
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 10
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 8
HEADACHE (Nervous system disorders) | 19 | 24
DYSGEUSIA (Nervous system disorders) | 9 | 7
DIZZINESS (Nervous system disorders) | 5 | 5
NEUROPATHY (Nervous system disorders) | 3 | 5
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 4
HYPOAESTHESIA (Nervous system disorders) | 4 | 2
RASH (Skin and subcutaneous tissue disorders) | 17 | 26
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 12
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 | 5
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 5
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 5
ACNE (Skin and subcutaneous tissue disorders) | 1 | 4
INSOMNIA (Psychiatric disorders) | 16 | 11
ANXIETY (Psychiatric disorders) | 12 | 7
DEPRESSION (Psychiatric disorders) | 10 | 7
URINARY TRACT INFECTION (Infections and infestations) | 16 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 4
CELLULITIS (Infections and infestations) | 5 | 1
SINUSITIS (Infections and infestations) | 0 | 4
DYSURIA (Renal and urinary disorders) | 13 | 6
MICTURITION URGENCY (Renal and urinary disorders) | 4 | 3
POLLAKIURIA (Renal and urinary disorders) | 6 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 4 | 2
HAEMATURIA (Renal and urinary disorders) | 5 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 4
FLUSHING (Vascular disorders) | 7 | 3
HOT FLUSH (Vascular disorders) | 6 | 2
HYPOTENSION (Vascular disorders) | 5 | 3
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 3 | 5
TACHYCARDIA (Cardiac disorders) | 4 | 3
VISION BLURRED (Eye disorders) | 3 | 5
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 3 | 5
CONTUSION (Injury, poisoning and procedural complications) | 4 | 3
HYPERSENSITIVITY (Immune system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.